CLINICAL TRIAL: NCT05020301
Title: Investigation of Functional Brain Network in Altered Meditation State With Multimodal Neuroimaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: School of Biomedical Engineering, Shanghai Jiao Tong University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: B20200361
Record Dates: First submitted 2021-07-14; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-06

CONDITIONS: Meditation; Mindfulness
Keywords: mindfulness; functional brain network; neuroimaging; meditation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Participants who have never practiced mindfulness
  Interventions: Device: external meditation guided audio; Device: internal meditation guided audio
- Beginner Practitioner (Experimental): Participants with less than two years of mindfulness practice
  Interventions: Device: external meditation guided audio; Device: internal meditation guided audio
- Advanced Practitioner (Experimental): Participants with more than two years of mindfulness practice
  Interventions: Device: external meditation guided audio; Device: internal meditation guided audio

INTERVENTIONS:
Device: external meditation guided audio — Examining DMN connectivity and CSF flow in external meditation state by External Meditation Instruction Audio.
Device: internal meditation guided audio — Examining DMN connectivity and CSF flow in external meditation state by Internal Meditation Instruction Audio.

SUMMARY:
The purpose of this study is to investigate functional brain network in altered meditation state with multimodal neuroimaging.

DETAILED DESCRIPTION:
1. Recruiting participants by approaching mindfulness training, poster, and websites.
2. Completing Questionnaires, Tests, and other materials for experiments.
3. Examining Functional Brain Network of Internal and External Meditation of practitioners with a meditation using multimodal neuroimaging.
4. Collecting and evaluating data about the connection of internal and external meditation with multimodal neuroimaging and identifying the function related to meditation state.

ELIGIBILITY:
Inclusion Criteria:

* A sufficient level of education to understand study procedure and be able to communicate with site personnel.
* 18-60 years old.
* Interested in meditation.
* No metal or electronic implants in the body; no prosthesis (metal braces, dentures, etc.); no claustrophobia; no tattoos, piercings, etc.; no makeup on the day of the experiment.
* Right-handed.

Exclusion Criteria:

* The participant has a contraindication to MRI examination, such as claustrophobia.
* The participant is physically unfit for MRI, such as having a metal implant.
* The participant has a history of neurological or psychiatric disorders, or is taking any chronic medications that may interfere with the experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Mindfulness positive awareness examined by Mindful Attention Awareness Scale (MAAS), Five Facet Mindfulness Questionnaire(FFMQ), The Chinese version of Freiburg Mindfulness Inventory(FMI-13) after the 1-week practice of internal and external mindfulness | Week 2
  MAAS is a validated, fifteen-item self-report measure on which the items are scored using a six-point rating scale (1 = almost always and 6 = almost never). The global score of the scale is obtained by calculating the mean score of each participant's responses, and higher scores on the scale convey the higher levels of dispositional mindfulness.
  FFMQ is a validated, self-administered questionnaire that measures the tendency to act with mindfulness. Its 39 items are assessed on a Likert scale from 1 to 5 (i.e., "never or very rarely true" to "very often or always true"). The higher scores on the scale convey the higher tendency to act with mindfulness.
  FMI-13 is a validated, thirteen-item self-report measure on which the items are scored using a four-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). This short form was used for measuring mindfulness traits, and higher scores on the scale convey the higher levels of mindfulness trait.
The mental states examined by Brief Profile of Mood States(Brief-POMS), Perceived Stress Scale(PSS) after the 1-week practice of internal and external mindfulness | Week 2
  The Brief-POMS is a validated,30-item measure, with items scored on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The scores for all items are pooled to generate a total score in the range of 0 to 120. A higher total score on the scale indicates a worse mood state.
  PSS is a validated, self-reported measure of psychological stress level. There are 10-items scored from 0 (never) to 4 (very often). The scores for all items are pooled to generate a total score in the range of 0 to 40. Higher total scores indicate the increasing level of psychological stress.
Cognitive impairment quantitative assessment by Mini-Mental State Examination(MMSE) | Week 2
  MMSE is a validated, widely used screening tool for cognitive impairment quantitative assessment. It included 11 items. The scores for all items are pooled to generate a total score in the range of 0 to 30. A 27-point was proved to be an appropriate cutoff for cognitive impairment in a population with relatively high educational attainment.
The cognitive flexibility examined by Cognitive Flexibility Inventory(CFI) after the 1-week practice of internal and external mindfulness | Week 2
  CFI is a validated, self-reported measure of cognitive flexibility，which consists of 20 statements scored from 1 ( "definitely disagree") to 7( "definitely agree."). The scores for all items are pooled to generate a total score of 20 to 140. Higher total scores indicate the increasing level of cognitive flexibility.
The ability of self-compassion examined by Self-Compassion Scale(SCS) after 1-week practice of internal and external mindfulness | Week 2
  SCS is a validated, 26-item self-report measure on which the items are scored using a five-point Likert scale scored from 1 (almost never) to 5 (almost always). The higher total score on the scale indicates a higher level of self-compassion.
Intelligence assessment by Raven's Standard Progressive Matrices (SPM) | Week 2
  SPM is a validated intelligence assessment that consists of 60 non-colored diagrammatic puzzles with a missing part, which subjects should correctly choose one among six options. SPM scores were estimated as the total of participants' correct answers (0-60). Higher total scores indicate the increasing level of intelligence level.
Mental flexibility assessment by Trail Making Test (TMT) | Week 2
  TMT is a validated mental flexibility assessment consisting of two parts (TMT-A and TMT-B ). The TMT-A consisted of a standardized page on which the numbers 1 to 25 were scattered within circles. The participants were asked to connect the numbers in order as quickly as possible. Similarly, the TMT-B consisted of a standardized page that included the numbers 1 to 13 and the letters A to L, which were randomly distributed. The participants were instructed to draw lines connecting numbers and letters (ascending and alphabetical) in alternating numbers and letters. A maximum time of 300 s was allowed before discontinuing the test. Direct scores of TMT were the time in seconds taken to complete each task (A and B). A Higher result indicates a worse cognitive outcome.
CSF pulsation index | Week 2
  CSF pulsation index, calculated by the number of CSF pulsation per minute.
Functional connectivity | Week 2
  Checking functional connectivity in major resting-state brain networks (such as DMN).

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Study Chair — Shanghai Mental Health Center; Jie Luo, Study Chair — School of Biomedical Engineering, Shanghai Jiao Tong University
Locations (1):
- School of Biomedical Engineering, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China